CLINICAL TRIAL: NCT01409785
Title: A Prospective, Randomized Comparison of the LMA Unique and LMA Supreme in Children
Brief Title: A Comparison of the LMA Unique and LMA Supreme in Children
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Narasimhan Jagannathan, Principal investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: LMA unique vs LMA supreme
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Children
Keywords: supraglottic airway devices in children

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- LMA Supreme
- LMA unique

SUMMARY:
The goal of this study is to compare the LMA Unique and LMA Supreme in children having surgery. We hypothesize that the airway leak pressures with the LMA Supreme will be superior to the LMA Unique. Airway leak pressures will be measured by recording the circuit pressure at which equilibrium is reached. The ease of placement, fiberoptic grade of laryngeal view, feasibility of use, and complications (airway related, gastric insufflation, trauma) will also be assessed.

DETAILED DESCRIPTION:
The LMA Supreme is a newer version of the current model, the laryngeal mask airway Unique. Both models are approved for use by the FDA, and are routinely used for airway management during general anesthesia. Three main features distinguish the laryngeal mask airway Supreme from the original LMA: i) a curved rigid airway tube, ii) provision for a gastric drain tube, and iii) a larger mask for improved fit and airway seal.

The aim of this randomized prospective study is to compare two types of the laryngeal mask airway: the laryngeal mask airway Unique and the laryngeal mask airway Supreme, in pediatric patients without the use of neuromuscular blockade. Based on the design features listed above, we hypothesize that the airway leak pressures with the LMA Supreme will be superior to the LMA Unique. Airway leak pressures will be measured by recording the circuit pressure at which equilibrium is reached. The ease of placement, fiberoptic grade of laryngeal view, feasibility of use, and complications (airway related, gastric insufflation, trauma) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing general anesthesia using a supraglottic airway device
* weight 10-25kg
* age 6 months-6 years

Exclusion Criteria:

ASA class IV, V Emergency procedures

* History of a difficult airway
* Active gastrointestinal reflux
* Active upper respiratory tract infection

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children weighing 10 to 25 kg undergoing surgical or medical procedures under anesthesia requiring a supraglottic airway device
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Airway leak pressure | after placement of the supraglottic airway device/ Participants will be followed 24 hours postoperatively
  Airway leak pressures will be measured by recording the circuit pressure at which equilibrium is reached when fresh gas flow is delivered at 3L/min when the pressure limiting valve is closed completely.

SECONDARY OUTCOMES:
Fiberoptic grade of laryngeal view | After placement of the supraglottic device
  The laryngeal alignment through the devices will be graded using an established scoring system
Adverse effects | Participants will be followed 24 hours postoperatively
  complications such as oxygen desaturations, mucosal trauma, reflex activation of the airway, sore throat, dysphonia will be recorded
Time to secure the airway | after placement of the supraglottic airway device
  From picking up the airway device to bilateral chest expansion and presence of ETCO2
Number of attempts to place the device | at the beginning of anesthesia
  number of attempts needed for successful placement will be recorde (maximum of 3 attempts will be considered as a failure)
Fiberoptic view through the gastric tube | After placement of the LMA supreme
  The view through the gastric drain tube of the LMA supreme will be assessed and graded using an established scoring system
Ease of gastric tube placement | After placement of the LMA supreme
  The ease of gastric placement will be assessed using a subjective scale
Gastric insufflation | During leak pressure testing
  The presence of gastric insufflations will be assessed during leak pressure testing by using epigastric auscultation
Quality of the airway | During maintenance of anesthesia
  The quality of hands free anesthesia will be assessed during maintenance of anesthesia using a previously described scale

CONTACTS AND LOCATIONS:
Overall Officials: narasimhan jagannathan, MD, Principal Investigator — childrens memorial hospital
Locations (1):
- Childrens Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Verghese C, Ramaswamy B. LMA-Supreme--a new single-use LMA with gastric access: a report on its clinical efficacy. Br J Anaesth. 2008 Sep;101(3):405-10. doi: 10.1093/bja/aen174. Epub 2008 Jun 17. PMID 18559351
- [Background] Timmermann A, Cremer S, Eich C, Kazmaier S, Brauer A, Graf BM, Russo SG. Prospective clinical and fiberoptic evaluation of the Supreme laryngeal mask airway. Anesthesiology. 2009 Feb;110(2):262-5. doi: 10.1097/ALN.0b013e3181942c4d. PMID 19194153
- [Background] Cook TM, Gatward JJ, Handel J, Hardy R, Thompson C, Srivastava R, Clarke PA. Evaluation of the LMA Supreme in 100 non-paralysed patients. Anaesthesia. 2009 May;64(5):555-62. doi: 10.1111/j.1365-2044.2008.05824.x. PMID 19413827
- [Background] White MC, Cook TM, Stoddart PA. A critique of elective pediatric supraglottic airway devices. Paediatr Anaesth. 2009 Jul;19 Suppl 1:55-65. doi: 10.1111/j.1460-9592.2009.02997.x. PMID 19572845